CLINICAL TRIAL: NCT00539097
Title: Evaluation Perioperative Nutrition on Donor Site Healing in Patients Undergoing Reconstructive Burn Surg
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: change in donor site care protocol; donor site healing is a study endpoint
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Theresa Mayes, Clinical Dietitian, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-04-23-05
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Burn; Reconstructive Surgical Procedure
Keywords: pediatrics
MeSH Terms: conditions — Burns

ARMS (2):
- A, treated (Experimental): treated with Juven po supplement x 3 weeks postop
  Interventions: Dietary Supplement: Juven (Ross Products) protein supplement
- B, control (No Intervention): Usual nutrition therapy received postop

INTERVENTIONS:
Dietary Supplement: Juven (Ross Products) protein supplement — Juven supplement oral x 3 weeks postop
  Arms: A, treated

SUMMARY:
The investigators hope to learn if taking a nutrition drink for a short time after surgery for an elective reconstructive burn injury improves donor site healing, muscle mass and scar maturation time (the point at which the redness, height and firmness of the wound has faded, flattened and softened, and no longer changes in appearance).

ELIGIBILITY:
Inclusion Criteria:

* At least one year post-acute burn injury
* Admitted for surgery whereby split thickness donor site created
* Received initial acute treatment at Shriner's Hospital in Cincinnati

Exclusion Criteria:

* Less than 6years of age
* Less than one year from acute burn injury
* Split thickness donor site/autograft not anticipated
* Initial treatment not at Shriners Hospital in Cincinnati

Ages: 6 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2005-06; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
donor site healing time | 3weeks

CONTACTS AND LOCATIONS:
Overall Officials: Theresa M Mayes, RD,LD, Principal Investigator — Shriners Hospital for Children, Cincinnati, Ohio
Locations (1):
- Shriners Hospital for Children, Cincinnati, Ohio, United States